CLINICAL TRIAL: NCT07301216
Title: Monitoring of Therapy in Wilson Disease With Off-Treatment Urinary Copper Excretion (OT-UCE): Comparison With Serum Non-Ceruloplasmin Copper (NCC) Assays
Brief Title: Off Treatment Urinary Copper Excretion in Wilson Disease, Pilot Study
Status: Recruiting | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2000040776; 1R01DK137861-01A1 (NIH)
Record Dates: First submitted 2025-12-22; First posted 2025-12-24 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Wilson Disease
Keywords: Urine copper excretion; Non-ceruloplasmin bound copper
MeSH Terms: conditions — Hepatolenticular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- OT-UCE and NCC for Zinc treated WD patients: OT-UCE and NCC will be measured in WD patients on Zinc therapy
- OT-UCE and NCC for Trientine treated WD patients: OT-UCE and NCC will be measured in WD patients on trientine therapy
- OT-UCE and NCC for Penicillamine treated WD patients: OT-UCE and NCC will be measured in WD patients on Penicillamine therapy

SUMMARY:
This is a prospective study that will determine the optimal timing for 24-hour urinary copper excretion (UCE) measurement after temporary discontinuation of standard therapies in Wilson Disease (WD) patients. The primary objective is to assess whether off-treatment UCE (OT-UCE) correlates with non-ceruloplasmin-bound copper (NCC) levels, aiming to validate OT-UCE as a surrogate marker for systemic copper bioavailability and disease stability. Stable WD patients will be enrolled, temporarily taken off treatment under close monitoring, and undergo UCE and NCC testing. If OT-UCE is validated, it could serve as a practical biomarker for monitoring WD treatment and stability in clinical practice and future trials.

DETAILED DESCRIPTION:
Study procedures will include providing multiple urine samples over a 24-hour period, storing the urine samples, and returning them during the end-of-study visit. Blood samples will be collected to measure copper levels and liver function. An in-person end-of-study visit will be attended.

Participation in this study will involve a brief stoppage of current Wilson Disease treatment.

Participants will perform 24-hour urine collections and communicate with study personnel daily during the brief time medication is not taken.

At the end-of-study visit, the investigators will collect urine samples, obtain blood samples, perform a physical exam, and review safety evaluations (communication with study personnel) made during the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Wilson Disease as defined by Leipzig score ≥4.
* Provision of signed and dated informed consent form.
* Stated willingness to comply with all study procedures (serial 24 h urine collections and local collection of samples for NCC, liver function and estimated GFR) and availability for the duration of the study.
* Treated WD for at least 12 months prior to study entry.
* Aminotransferase values (ASAT and ALAT) < 2 times the upper limit of normal (ULN).
* INR < 1.5 or stable INR for those with initial elevated INR for at least six months prior to study entry in the absence of anticoagulation therapy.
* Renal function defined as eGFR > 30 cc/min.
* No change of WD therapy during the previous 6 months of study enrollment.

Exclusion Criteria:

* Current dual / mixed therapy for WD (i.e. zinc and d-penicillamine or trientine at the same time)
* Current Pregnancy or lactation. *
* Recent estrogen-based treatment (in the last month).
* Cirrhosis with recent hepatic decompensation (within the last 6 months) - new onset of ascites, spontaneous bacterial peritonitis, esophageal variceal bleeding, or hepatic encephalopathy
* Investigator believes the patient will be unable to do the required 24-hour urine studies and participate in the follow up visits as expected.
* Previous non-compliance for therapy and/or to low-copper diet that would compromise the evaluation of previous UCE and/ or results from the off-treatment period.

  * Childbearing aged patients recruited outside of the registry will be reviewed, and the patients will be asked to perform an initial urine pregnancy test prior to the recommended blood testing (approximately 60 to 90 days prior to intervention). They will be permitted to continue with the screening process if the result is negative. They will be asked to perform a second urine pregnancy test as close as possible prior to study intervention (discontinuation of treatment). If the result of the second pregnancy test is negative they will be permitted to continue with the protocol, but if the result is positive they will be excluded from further participation at that time.

Childbearing aged patients recruited from the registry who meet inclusion criteria and may move directly to the study intervention will be required to perform a urine pregnancy test as close as possible to the time prior to the initiation of the study protocol (discontinuation of treatment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with confirmed Wilson Disease (Leipzig score ≥4), and stable disease will be screened and recruited for this pilot. This will include patients 18 years old and above as the intervention for this study is a temporary discontinuation of therapy, and this group of patients will tolerate this intervention with minimal risk.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Mean concentration of OT-UCE for each standard of care WD treatment | days 1, 2, 3 and 4 post stopping WD meds
  Urine samples will be collected daily for 4 days after stopping WD medications. The sequential evaluation of OT-UCE over a maximum of 4 days after treatment withdrawal will allow investigators to define the optimal ranges for UCE and select the best time-point for OT-UCE evaluations for WD patients on the 3 different therapies.
Mean NCC concentration for each WD treatment | days 1, 2, 3 and 4 post stopping WD meds
  Measure NCC and assess the correlation between NCC and OT-UCE Urine samples will be collected daily for 4 days after stopping WD medications. The sequential evaluation of NCC over a maximum of 4 days after treatment withdrawal will allow investigators to assess the correlation between NCC and OT-UCE.

SECONDARY OUTCOMES:
Mean OT-UCE Ranges for each WD med | days 1, 2, 3 and 4 post stopping WD meds
  Urine samples will be collected daily for 4 days after stopping WD medications. The sequential evaluation of OT-UCE over a maximum of 4 days after treatment withdrawal will allow investigators to define the optimal ranges for UCE for WD patients on the 3 different therapies.
Assess the best timepoints for performance of OT-UCE for each drug | days 1, 2, 3 and 4 post stopping WD meds
  The day (or the minimal number of consecutive days) after treatment interruption at which 24-hour OT-UCE stabilizes (defined as a plateau with less than 10% variability between two consecutive measurements) for each drug (zinc, penicillamine, trientine). This will define the optimal timing of OT-UCE monitoring for each treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Michael L Schilsky, MD FAASLD, Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Solovyev N, Ala A, Schilsky M, Mills C, Willis K, Harrington CF. Biomedical copper speciation in relation to Wilson's disease using strong anion exchange chromatography coupled to triple quadrupole inductively coupled plasma mass spectrometry. Anal Chim Acta. 2020 Feb 15;1098:27-36. doi: 10.1016/j.aca.2019.11.033. Epub 2019 Nov 15. PMID 31948584
- [Background] Harrington CF, Carpenter G, Coverdale JPC, Douglas L, Mills C, Willis K, Schilsky ML. Accurate non-ceruloplasmin bound copper: a new biomarker for the assessment and monitoring of Wilson disease patients using HPLC coupled to ICP-MS/MS. Clin Chem Lab Med. 2024 Jul 30. doi: 10.1515/cclm-2024-0213. Online ahead of print. PMID 39072400